CLINICAL TRIAL: NCT06814834
Title: A Prospective Study to Compare the Efficacy of Oral Dissolution Therapy (ODT), Extracorporeal Shock Wave Lithotripsy (ESWL), and Combined ESWL and ODT as Non-Invasive Modalities for Treating Small and Medium-Sized Radiolucent Renal Stones
Brief Title: The Efficacy of Oral Dissolution Therapy (ODT), Extracorporeal Shock Wave Lithotripsy (ESWL), and Combined ESWL and ODT as Non-Invasive Modalities for Treating Small and Medium-Sized Radiolucent Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ateya, Lecturer of Urology, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-556-2023
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Oral Dissolution Therapy; Extracorporeal Shock Wave Lithotripsy; Noninvasive; Small; Medium; Radiolucent Renal Stones
MeSH Terms: conditions — Cerebral Palsy | interventions — Lithotripsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral dissolution therapy group (Active Comparator): Patients received guidance for oral potassium-sodium-hydrogen-citrate (6:6:3:5) at a dosage of twenty milliequivalents three times every day, along with a daily fluid intake of two to three liters and a food plan to restrict protein and sodium consumption for a maximum of three months.
  Interventions: Drug: Oral dissolution therapy
- Extracorporeal shock wave lithotripsy group (Experimental): Patients received extracorporeal shock wave lithotripsy utilizing a Dornier lithotripter equipped with an integrated ultrasound for stone localization. If the patient required additional sessions, up to a maximum of four sessions, at a rate of 60-90 shocks per minute, the period between sessions was three weeks.
  Interventions: Procedure: Extracorporeal shock wave lithotripsy
- Oral dissolution therapy + extracorporeal shock wave lithotripsy group (Experimental): Patients received a combination of oral dissolution therapy and extracorporeal shock wave lithotripsy.
  Interventions: Procedure: Oral dissolution therapy + extracorporeal shock wave lithotripsy

INTERVENTIONS:
Drug: Oral dissolution therapy — Patients received guidance for oral potassium-sodium-hydrogen-citrate (6:6:3:5) at a dosage of twenty milliequivalents three times every day, along with a daily fluid intake of two to three liters and a food plan to restrict protein and sodium consumption for a maximum of three months.
  Arms: Oral dissolution therapy group
Procedure: Extracorporeal shock wave lithotripsy — Patients received extracorporeal shock wave lithotripsy utilizing a Dornier lithotripter equipped with an integrated ultrasound for stone localization. If the patient required additional sessions, up to a maximum of four sessions, at a rate of 60-90 shocks per minute, the period between sessions was three weeks.
  Arms: Extracorporeal shock wave lithotripsy group
Procedure: Oral dissolution therapy + extracorporeal shock wave lithotripsy — Patients received a combination of oral dissolution therapy and extracorporeal shock wave lithotripsy.
  Arms: Oral dissolution therapy + extracorporeal shock wave lithotripsy group

SUMMARY:
This study aimed to compare oral dissolution therapy (ODT), extracorporeal shock wave lithotripsy (ESWL), and a combination of ESWL and ODT as noninvasive modalities for treating small and medium-sized renal radiolucent.

DETAILED DESCRIPTION:
Various methods exist for managing small and medium-sized radiolucent renal stones. These range from observation to oral dissolution therapy (ODT), percutaneous nephrolithotomy (PCNL), retrograde intrarenal surgery (RIRS), and extracorporeal shock wave lithotripsy (ESWL).

Oral dissolving therapy diminishes the recurrence rates of stones. It positively influences the medical management of stone activity following ESWL in cases with residual calculi. By integrating oral dissolution therapy with extracorporeal shock wave lithotripsy, cases may experience the advantages of both non-invasive techniques. The combination of oral dissolution therapy and ESWL is an efficient therapeutic modality for radiolucent renal stones, dramatically reducing the overall stone volume. It also reduces the frequency of necessary extracorporeal shock wave lithotripsy sessions compared to treatment with ESWL alone

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Patients with a single radiolucent renal stone 0.5-2 cm at largest diameter diagnosed by non-contrast MSCT of the urinary tract (CTUT) ≤ 500 HU (Hounsfield Unit) and not seen on kidney, ureter, and bladder (KUB) X-ray.

Exclusion Criteria:

* Patients with Coagulation disorders, a pacemaker, severe deformity of the skeletal system, anatomical obstruction distal to the stone, and obesity (Body Mass Index more than or equal to 35 kilograms per meter square).
* Patients with renal insufficiency (creatinine more than 1.7 mg/dl).
* Patients with active urinary tract infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Stone-free status | 3 months after the procedure
  To assess the stone-free status, which is characterized by no evidence of any residual stones in renal units by MSCT of the urinary tract (CTUT) at 3 months following oral dissolution therapy (ODT), extracorporeal shock wave lithotripsy (ESWL), or combined ODT and ESWL.

SECONDARY OUTCOMES:
Complication rate | 3 months after the procedure
  The complication rate of extracorporeal shock wave lithotripsy (ESWL) as hematuria, perinephric hematoma, renal colics, steinstrasse fragments, gastrointestinal tract upset, number of sessions needed, and the essential for auxiliary processes following 3 months as ureteroscopy (URS), Flexible URS, or percutaneous nephrolithotomy (PCNL).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.